CLINICAL TRIAL: NCT03302364
Title: A Research in Pharmacogenomics and Accurate Medication of Risperidone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of Pharmacy,M.D.& Ph.D., Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2016[1240]
Record Dates: First submitted 2017-09-27; First posted 2017-10-05 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Mental Illness
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Risperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples With DNA — Whole blood samples will be drawn and collected, serum sample will also be obtained by centrifugation of whole blood at 4 ℃. The collected samples will be further detected and the concentration data will be used for PG-PK, PG-PD and PG-ADR analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- risperidone patients: patients that are in accordance with DSM-IV-TR schizophrenia diagnostic criteria, based on concise International Neuropsychological Interview(MINI)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — patients who have never received risperidone or who have received re-administration of risperidone after discontinuation of risperidone treatment
  Other Names: Risperidal

SUMMARY:
Risperidone is a selective monoamine receptor antagonist. It plays an antipsychotic effect by antagonizing 5-HT2 / D2 receptor. As a second-generation antipsychotic drug, risperidone is metabolized to 9-hydroxy Risperidone in the body very quickly. There are individual differences in the pharmacokinetics and pharmacodynamics of risperidone. For example, CYP2D6 genotype can greatly affect the metabolism of risperidone, and provide evidence for adjusting the type and dose of medication to treat Schizophrenia. In this study, we will verify the correlation between the polymorphisms of genes related with risperidone drug metabolites, drug transporters, drug targets and drug metabolism, pharmacodynamics, adverse reactions in Chinese population, providing basis for clinical rational use of risperidone.

DETAILED DESCRIPTION:
Subjects with schizophrenia will be recuited from several sub-centers. The relevant gene polymorphisms and risperidone drug metabolism, drug adverse reaction parameters are monitored through drawing blood samples at 0h, 6h, D27 and D56 of the risperidone drug administration. Information related to drug pharmacokinetics, pharmacodynamics and adverse reactions(serum prolactin levels) will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients that meet with DSM-IV-TR schizophrenia diagnostic criteria, based on concise International Neuropsychiatric Interview (MINI);
* patients who have never received risperidone treatment or who need re-administration of risperidone after previous treatment with risperidone;
* Subjects and / or their guardians who agree to sign the informed consent.

Exclusion Criteria:

* patients who use CYP2D6 or CYP3A4 inducers or inhibitors as treatment drugs;
* patients with hepatic insufficiency;
* patients with renal insufficiency;
* patients who use other drugs that interact with risperidone;
* certain patients that the researchers consider to be unsuitable for the clinical trail.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Schizophrenic patients who are going to be treated with risperidone.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-10-22 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
genotype | Pre-dose of risperidone
  The genotypes of subjects are detected.

SECONDARY OUTCOMES:
Prolactin concentration in plasma | Hour 0, Weeks 6-8
  Prolactin concentration is determined by ELISA method, it is one of the ADR of prolactin.
risperidone and 9-OH-risperidone concentration in plasma | day 1,day 2
  Risperidone and 9-OH-risperidone concentration are PK outcomes for evaluation.
Negative and positive scale | day-1,day28±2，day56±2
  PANSS scole of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, Ph.D & M.D, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China